CLINICAL TRIAL: NCT04290676
Title: DEXYCU (Dexamethasone Intraocular Suspension) 9% Retrospective Study 001
Acronym: DEXYCURetro
Status: Completed | Type: Observational
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DEXYCU Retrospective Study 001
Record Dates: First submitted 2019-11-27; First posted 2020-03-02 (Actual); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Cataract
Keywords: DEXYCU; Cataract; dexamethasone intraocular suspension
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DEXYCU (dexamethasone intraocular suspension) 9%.: DEXYCU (dexamethasone intraocular suspension) 9%. Single dose, intraocularly in the posterior chamber at the end of surgery. The dose is 0.005 mL of dexamethasone 9% (equivalent to 517 micrograms).
  Interventions: Drug: DEXYCU (dexamethasone intraocular suspension) 9%.

INTERVENTIONS:
Drug: DEXYCU (dexamethasone intraocular suspension) 9%. — DEXYCU contains dexamethasone 9% w/w (103.4 mg/mL) as a sterile suspension for intraocular ophthalmic administration. DEXYCU is provided as a kit for administration of a single dose of 0.005 mL of 9% dexamethasone (equivalent to 517 micrograms of dexamethasone).
  Other Names: dexamethasone intraocular suspension

SUMMARY:
Retrospective study to provide clinical outcomes with DEXYCU (dexamethasone intraocular suspension) 9%.

DETAILED DESCRIPTION:
This retrospective study is intended to provide large-scale, real-world data on clinical outcomes with DEXYCU (dexamethasone intraocular suspension) 9%.

ELIGIBILITY:
Inclusion Criteria

* Male and Female subjects at least 18 years of age
* Subjects who underwent cataract surgery from 12Mar2019 to 15Dec2019 and received DEXYCU

Exclusion Criteria

• Subjects who underwent cataract surgery and did not receive DEXYCU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent cataract surgery from 12Mar2019 to 15Dec2019 and received DEXYCU
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dario Paggiarino, MD, Principal Investigator — Senior Vice President, Chief Medical Officer, EyePoint Pharmaceuticals; Keyur Patel, PharmD, Study Chair — Vice President, Medical Affairs, EyePoint Pharmaceuticals; Flavio Leonin, Jr., MD, Study Director — Senior Manager, Clinical Affairs, EyePoint Pharmaceuticals
Locations (22):
- United States (22):
  - Eye Center South Locations, Dothan, Alabama
  - Inland Eye Specialists, Hemet, California
  - Harvard Eye Associates, Laguna Hills, California
  - Coastal Vision Medical Group, Orange, California
  - North Bay Eye Associates, Inc., Rohnert Park, California
  - The Eye Associates of Manatee, LLP, Bradenton, Florida
  - Eye Physicians of Pinellas, PA, dba The Eye Institute of West Florida, Largo, Florida
  - Jacksoneye, SC, Lake Villa, Illinois
  - Hauser-Ross Eye Institute, Oak Brook, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - Physicians Eyecare Center, Baltimore, Maryland
  - Discover Vision Centers, Independence, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Surgery Center of Central New Jersey, Pennington, New Jersey
  - SightMD, PLLC, Hauppauge, New York
  - New York Eye Surgery Center, The Bronx, New York
  - Island Eye Surgicenter, Westbury, New York
  - Wills Surgery Center, Jenkintown, Pennsylvania
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Valley Retina Institute, PA, McAllen, Texas
  - The Eye Centers of Racine and Kenosha, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- DEXYCU (Dexamethasone Intraocular Suspension) 9%: All participants received DEXYCU (dexamethasone intraocular suspension) 9% as a single dose, administered intraocularly into the posterior chamber at the end of surgery.
Period: Overall Study
Arm/Group | DEXYCU (Dexamethasone Intraocular Suspension) 9%
Started | 527; 641 eyes
Completed | 527; 641 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | DEXYCU (Dexamethasone Intraocular Suspension) 9%
Number analyzed (Participants) | 527
Number analyzed (eyes) | 641
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308
  Male | 219
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 74
  Ethnicity: Not Hispanic or Latino | 327
  Ethnicity: Not Reported | 100
  Ethnicity: Unknown | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Anterior Chamber Cell Grade 0
Description: Of eyes with a record at postoperative day 8, percentage with anterior chamber cell grade 0. Cells in the anterior chamber of the eye are indicative of intraocular inflammation and are evaluated using a slit-lamp biomicroscope; a grade of 0 indicates that no inflammatory cells were visible in a 1 mm by 1 mm slit beam.
Time Frame: Postoperative day 8
Population: eyes with a record at postoperative day 8
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | DEXYCU (Dexamethasone Intraocular Suspension) 9%
Number analyzed (Participants) | 315
Number analyzed (eyes) | 315
percentage of eyes | 65

ADVERSE EVENTS:
Time Frame: This was a retrospective observational study based on chart review of patients in real-world clinical settings receiving DEXYCU after cataract surgery between 12 March and 15 December 2019. Data from patient charts were entered retrospectively by the study coordinator or other designated, trained personnel at study sites into a password-protected database, for the day of surgery and for postoperative days 1, 8, 14, and 30, as available.
Description: All adverse events reported by investigators are included, irrespective of whether or not the event was present prior to intraocular administration of DEXYCU at the end of cataract surgery.
Arm/Group | DEXYCU (Dexamethasone Intraocular Suspension) 9%
All-Cause Mortality (participants affected / at risk) | 0/527
Serious Adverse Events (participants affected / at risk) | 0/527
Other Adverse Events (participants affected / at risk) | 20/527
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEXYCU (Dexamethasone Intraocular Suspension) 9% (N=527)
Intraocular pressure increased (Investigations) | 6 (7)
Corneal edema (Eye disorders) | 5 (6)
Iritis (Eye disorders) | 4 (4)
DEXYCU on lens optic (Product Issues) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Retina peripheral hole (Eye disorders) | 1 (1)
Hypotony maculopathy (Eye disorders) | 1 (1)
Retained cortex in anterior chamber (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
During the Study and for a period of ten (10) years after completion or early termination of the Multi-Center Retrospective Trial, without Sponsor's and/or its representative prior written consent, Institution and Investigator will not publish, disseminate or otherwise disclose, deliver or make available any Confidential Information to any third party other than Study Personnel or Sponsor's representative, and then only for the purpose of conducting the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04290676/Prot_SAP_000.pdf